CLINICAL TRIAL: NCT04612673
Title: Anti-PD-1 Antibody, Sintilimab, as Second-line Therapy for Advanced or Metastatic Non-small Cell Lung Cancer Patients : a Phase II, Historical Control, Biomarker-selected Study
Brief Title: A Phase II Study of Anti-PD-1 Antibody, Sintilimab, as Second-line Therapy for Biomarker-selected Advanced or Metastatic NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Medical University, China (Other)
Collaborators: Shengjing Hospital (Other); The First People's Hospital of Jingzhou (Other); The People's Hospital of Liaoning Province (Other); Liaoning Cancer Hospital & Institute (Other); Anshan Tumor Hospital (Other); Benxi Cental Hospital (Other); The Second Affiliated Hospital of Dalian Medical University (Other); The First Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Principal Investigator, Yunpeng Liu, Director of Department of Medical Oncology, China Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI308Y035
Record Dates: First submitted 2020-10-28; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Participants received Sintilimab, 200mg, iv, d1, Q3W,and it should be continued until disease progress or toxicity cannot be tolerated or patients withdraw consent
  Interventions: Drug: Sintilimab

INTERVENTIONS:
Drug: Sintilimab — immune checkpoint inhibitor, 200mg, iv, d1,Q3W

SUMMARY:
The purpose of this study is to to explore the efficacy and safety of PD-1 immune check point inhibitor, sintilimab, in biomarker-selected subjects with advanced or metastatic Non-small Cell Lung Cancer who have failed from standard front-line treatment.

DETAILED DESCRIPTION:
This study is planned to be carried out in The First Hospital of China Medical University. 33 cases are preliminarily expected to be included. The study started in October 2020 and ended in October 2023. It is expected that the trial will end in October 2023.

In the absence of such situations as withdrawal of informed consent, intolerance of drug toxicity and side effects, or inappropriateness for further trials, each participant's expected time for research and treatment will continue until radiographically confirmed tumor progression occurs.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 and ≤ 70 years of age , regardless of gender；
* Pathologically confirmed diagnosis of locally advanced or metastatic NSCLC (according to the eighth edition of AJCC staging, IIIB, IIIC, IV), with at least one measurable lesion (RECIST 1.1)
* treatment failure after first-line standard treatment (definition of treatment failure: intolerable side effects, disease progression during or after treatment);
* No known EGFR sensitive mutations and ALK gene rearrangements.
* Tumor tissue samples that meet the testing requirements for biomarker testing can be provided. Testing will be carried out in the central laboratory.
* NSCLC that is anti-programmed cell death ligand 1 (PD-L1) positive(TPS PD-L1 expression is ≥1% ), and CD8 expression is ≥20% (pre-treatment samples are sufficient).
* ECOG PS: 0-1
* Sufficient organ and bone marrow function as defined below:

  1. Routine blood examination:

     1. HB≥90g/L;
     2. ANC ≥1.5×109/L;
     3. PLT ≥90×109/L;
  2. Biochemical inspection shall:

     1. Total bilirubin ≤ 1.5 ULN;
     2. ALT and AST≤2.5ULN;
     3. Serum Cr≤1ULN, endogenous creatinine clearance rate>60ml/min (Cockcroft-Gault);
* The international normalized ratio (INR) ≤ 1.5 and partial prothrombin time (PPT or APTT) ≤ 1.5 ULN within the 7 days before enrollment.
* Life span expectation over 3 months;
* Provide written informed consent;

Exclusion Criteria:

* Allergic to any ingredients of Sintilimab preparations; or have had severe allergic reactions to other monoclonal antibodies in the past.
* Received more than one regimen for the treatment of locally advanced or metastatic NSCLC in the past (except for adjuvant/neoadjuvant chemotherapy that has exceeded the 24-week).
* Received any anti-PD-1/PD-L1 antibody, anti-CTLA4 antibody, or other immunotherapy in the past.
* Diagnosed other malignant tumors within 5 years before the first administration, excluding radically cured skin basal cell carcinoma, skin squamous cell carcinoma and/or radically excised carcinoma in situ.
* Be treated with anti-tumor vaccines or other immunostimulatory anti-tumor drugs (interferon, interleukin, thymosin, immune cell therapy, etc.) within 1 month before enrolled.
* Central nervous system metastasis with symptoms..
* Acute or chronic active hepatitis B (defined as positive for hepatitis B virus surface antigen HBsAg during the screening period) or hepatitis C infection.
* History of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, drug-related pneumonia, severely impaired lung function and other lung diseases.
* Active tuberculosis (TB), who are receiving anti-tuberculosis treatment or have received anti-tuberculosis treatment within 1 year before the first administration.
* People infected with human immunodeficiency virus (HIV) (HIV antibody positive), people with known syphilis infection.
* Patients who are considered to be at greater medical risk due to severe, uncontrollable diseases, non-metastatic systemic diseases, or active, uncontrollable infections.
* An active autoimmune disease that requires systemic treatment (such as the use
* disease-relieving drugs, corticosteroids, or immunosuppressive agents) occurred within 2 years before the first administration.
* Have used immunosuppressive drugs within 4 weeks before the first administration, excluding nasal spray, inhaled or other local glucocorticoids or physiological doses of systemic glucocorticoids (ie not more than 10 mg/day prednisone Loose or equivalent doses of other glucocorticoids), allowing temporary use of glucocorticoids for the treatment of asthma, chronic obstructive pulmonary disease and other diseases such as dyspnea symptoms.
* Exclude subjects who are expected to require any other form of anti-tumor therapy (including maintenance therapy with other NSCLC drugs, radiotherapy, and/or surgical resection) in the study.
* Exclude those who underwent major surgery within 4 weeks before the first medication, those with non-thoracic radiation therapy >30 Gy within 4 weeks before the first medication, those with chest radiation >30 Gy within 24 weeks before the first medication, and 2 before the first medication Subjects who received palliative radiation <30 Gy within a week and who failed to recover from the toxicity and/or complications of these interventions to NCI-CTC AE ≤ 1 degree (except for hair loss and fatigue). Palliative radiotherapy for symptom control is permitted and must be completed at least 2 weeks before the start of treatment with the study drug, and there are no plans for additional radiotherapy to the same lesion. For patients who received radiotherapy 2 weeks before the first administration, all of the following conditions must be met before they can be enrolled: There is no radiotherapy-related toxic reaction, glucocorticoids are not required, and radiation pneumonitis, radiation hepatitis, radioactivity are excluded Enteritis and so on.
* Pregnancy or lactation.
* Participated in other drug clinical trials within four weeks.
* The investigator believes that there are any conditions that may damage the subject or result in the subject not being able to meet or perform the research request.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2020-11-20 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Progress free survival (PFS) | untill Progressive Disease(PD) or death(up to 24 months)
  PFS defined as the time from first dose of study treatment until the first date of either objective disease progression or death due to any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | From randomization until death (up to 24 months)
  OS is defined as the time until death due to any cause.
Objective Response Rate (ORR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  ORR is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1.prior to progression or any further therapy.
Disease Control Rate (DCR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Defined as the proportion of patients with a documented complete response, partial response, and stable disease (CR + PR + SD) based on RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Yunpeng Liu, PhD, Principal Investigator — China Medical University, China
Locations (1):
- The First Affiliated Hospital of China Medical University, Shenyang, Liaoning, China